CLINICAL TRIAL: NCT00367588
Title: Low Bacterial Diet in Patients With Cytopenia After Intensive Chemotherapy for Hematological Malignancy: a Study of Efficacy
Brief Title: Low Bacterial Diet in Patients With Cytopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TN3 / CvZ nr.01111
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2004-06

CONDITIONS: Cytopenia
Keywords: chemotherapy; diet; hematological malignancy; infection prevention; protective isolation; Patients with cytopenia due to intensive chemotherapy for hematological malignancy
MeSH Terms: conditions — Cytopenia; Hematologic Neoplasms

INTERVENTIONS:
Behavioral: Low bacterial diet

SUMMARY:
The purpose of this prospective, randomized study was to determine the efficacy of low bacterial diet, in comparison to normal hospital diet, with gut colonization by aerobic Gram negative rods and yeasts as primary endpoint. In addition, the occurrence of infections and the total costs of hospital care were documented, in order to identify potential cost savings by the use of either diet.

DETAILED DESCRIPTION:
Patients with hematological malignancies who receive intensive chemotherapy usually develop a period of cytopenia, during which there is an increased risk of infection. Mucositis can also develop in these patients, enabling micro-organisms, belonging to the endogenous intestinal flora, to translocate from the intestine to the lymphoid tissue and blood. Therefore, when mucositis and cytopenia develop simultaneously, the risk of infection increases further. In this regard bloodstream infection by Gram negative rods and yeasts are an important cause of serious infections causing considerable morbidity.

In order to reduce the risk of infection several preventive measures have been adopted. Fundamentally, all of these measures were designed to prevent either acquisition of Gram negative rods or fungal pathogens from the environment, or the translocation of these potential pathogens across the mucosal barrier of the gut. These measures include protective (or reverse) isolation, antibiotic prophylaxis with antibiotics which selectively eradicate the aerobic Gram negative rods and yeasts from the gut flora, and finally the use of low-bacterial diets.

In this prospective, randomized study on the efficacy of low bacterial diet, in comparison to normal hospital diet, gut colonization by aerobic Gram negative rods and yeasts, the occurrence of infections and the total costs of hospital care were chosen as study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* acute leukemia receiving remission induction chemotherapy
* receiving antibiotic prophylaxis for cytopenia leukocytes lower than 1000/mm3 in peripheral blood)
* informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Study Completion 2004-06

PRIMARY OUTCOMES:
Colonization of the gut by aerobic Gram negative rods and yeasts

SECONDARY OUTCOMES:
The occurrence of infections
The total societal costs

CONTACTS AND LOCATIONS:
Overall Officials: Frank H. van Tiel, MD, PhD, Principal Investigator — University Hospital Maastricht, Maastricht, the Netherlands
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands